CLINICAL TRIAL: NCT05419349
Title: Novel Staging Schemes for Siewert Type II Esophagogastric Junction Adenocarcinoma: A Real-World Data Cohort Study From SEER Database
Status: Completed | Type: Observational
Sponsor: Fujian Medical University Union Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: SEEREGJ-01
Record Dates: First submitted 2022-06-13; First posted 2022-06-15 (Actual); Last update posted 2022-11-04 (Actual); Status verified 2022-06

CONDITIONS: Adenocarcinoma of the Esophagogastric Junction
Keywords: esophagogastric junction; total examined lymph nodes; staging

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Procedure: esophagogastric junction cancer surgery — esophagogastric junction cancer surgery

SUMMARY:
This study have two aims, the first is to explore the optimal cutoff of TLN for Siewert type II AEG using the Surveillance, Epidemiology, and End Results (SEER) database the second is to provide a more accurate staging for Siewert type II AEG patients.

ELIGIBILITY:
Inclusion Criteria:

Siewert type for adenocarcinoma of the esophagogastric junction; pathologically confirmed T1-4aN0-3M0 stage after surgery after a pathological examination of the LNs.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: The data were obtained from the SEER public database. In the 18 SEER registries, the 2021 release of the public use dataset from 2004 to 2015 was queried.
Sampling Method: Non-Probability Sample
Enrollment: 1819 (Actual)
Dates: Start 2022-06-01 (Actual); Primary Completion 2022-06-07 (Actual); Study Completion 2022-06-07 (Actual)

PRIMARY OUTCOMES:
Overall survival | 5-year overall survival
  the time from disease diagnosis to death from any cause

CONTACTS AND LOCATIONS:
Locations (1):
- Fujian Medical University Union Hospital, Fuzhou, Fujian, China

IPD SHARING:
Plan to Share IPD: No
The data were obtained from the SEER public database